CLINICAL TRIAL: NCT05413148
Title: The Effect of Wharton Jelly-derived Mesenchymal Stem Cells and Stem Cell Exosomes on Visual Functions in Patients With Retinitis Pigmentosa
Brief Title: The Effect of Stem Cells and Stem Cell Exosomes on Visual Functions in Patients With Retinitis Pigmentosa
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Kuddusi Erkılıç, Principal Investigator, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TSG-2021-11599.
Record Dates: First submitted 2022-05-28; First posted 2022-06-09 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Retinitis Pigmentosa
Keywords: wharton jelly derived; mesenchymal stem cell; exosome
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wharton jelly-derived mesenchymal stem cell (Active Comparator): Single subtenon injection of Wharton jelly-derived mesenchymal stem cells will be performed on a single eye after randomization
  Interventions: Biological: Subtenon injection of Wharton jelly derived mesenchymal stem cells
- Mesenchymal stem cell exosome (Wharton jelly-derived) (Active Comparator): Single subtenon injection of mesenchymal stem cell exosomes (Wharton jelly-derived)will be performed on a single eye after randomization.
  Interventions: Biological: Subtenon injection of Wharton jelly derived mesenchymal stem cell exosomes
- Placebo (Placebo Comparator): A single subtenon injection of saline will be performed on a single eye after randomization.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Subtenon injection of Wharton jelly derived mesenchymal stem cells — Single subtenon's injection for single eye
  Arms: Wharton jelly-derived mesenchymal stem cell
Biological: Subtenon injection of Wharton jelly derived mesenchymal stem cell exosomes — Single subtenon's injection for single eye
  Arms: Mesenchymal stem cell exosome (Wharton jelly-derived)
Other: Placebo — Single Subtenon injection of saline for a single eye
  Arms: Placebo

SUMMARY:
This clinical trial aims to study the efficacy of umbilical cord-derived mesenchymal stem cells and their exosomes in the treatment of retinitis pigmentosa. The participants will be randomized into 3 groups. Functional and structural parameters will be compared before and after the injections and also will be compared among the groups to reveal whether stem cell and their exosomes are more effective than placebo.

DETAILED DESCRIPTION:
Retinitis pigmentosa (RP) is one of the leading causes of vision loss and irreversible blindness. It is stated that 1.4 million people are affected in the world and its prevalence is 1:4000. Stem cell applications are methods that are increasingly gaining importance in the field of regenerative medicine and ophthalmology. In addition to many experimental studies in retinal diseases including retinitis pigmentosa, there are also clinical studies reporting successful results on humans. The most widely used stem-cell group in current clinical practice is mesenchymal stem cells. The advantages are that they are relatively easy to obtain and do not induce severe immune responses. Clinical studies in stem cell therapies for the eye suggest that stem cells benefit the surrounding tissue by secreting support such as growth factors, and extracellular vesicles, mostly due to their trophic and paracrine effects. In intraocular applications, there has been a tendency to apply mesenchymal stem cells around/outside the eye, including subtenon and suprachoroidal application due to side effects such as retinal detachment and epiretinal membrane.

Other cellular products that have been studied in animal studies and clinical research in recent years are exosomes. Exosomes are a subgroup of extracellular vesicles released from cells. Exosomes are extracellular vesicles 30-150 nm in size and carry at least one of the exosomal proteins CD63, CD9, CD81, syntenin-1 and TSG101. Exosomes are secreted from different cells in the organism and are also found in body fluids. Exosomes play a role in the transportation of biomolecules such as lipids, carbohydrates, nucleic acids and proteins from one cell to another and in this way, they function in genetic information transfer, and reprogramming of the opposite cell and intercellular communication. One of the sources of exosomes is mesenchymal stem cells that secrete high amount of exosomes. Mesenchymal stem cell-derived exosomes have been reported to have therapeutic effects, just like mesenchymal stem cells. It is thought that stem cells also exert their clinical effects through paracrine factors they secrete rather than being implanted in the tissue. However, the mechanism of action of mesenchymal stem cells has not been fully understood, and exosomes are thought to contribute to the effect. The storage and durability of exosomes may provide advantages in therapeutic applications compared to mesenchymal stem cells and may provide more immunological advantages in allogeneic applications compared to cellular treatments since they do not contain cells.

One of the sources from which mesenchymal stem cells can be obtained is Wharton jelly, which is the mesenchymal tissue of the umbilical cord. Stem cells originating from Wharton gel are a good source of stem cells due to their high differentiation capacity, high regeneration capacity, constant doubling time, high proliferation capacity, low immunogenicity, and no ethical problems due to non-invasive methods, and easy availability.

This clinical trial will enroll patients diagnosed with retinitis pigmentosa. The diagnosis of RP is made by clinical fundus examination, examinations in our clinic, and genetic analysis.

At the beginning of the study, all volunteers will undergo a full ophthalmologic examination including best-corrected visual acuity, anterior segment and fundus examination with a slit lamp, OCT (optical coherence tomography), VF (visual field), ERG (electroretinogram), mfERG (multifocal ERG), OCTA (optical coherence tomography). Retinal and choroidal thickness and ellipsoid bandwidth in OCT, MD (mean deviation) value showing sensitivity in VF, amplitude and latency times in ERG and mf-ERG, vascular density and vascular flow ratios in OCTA will be recorded.

The volunteers will be randomized into three. The 1st group will be the placebo group (45 volunteers) and 0.5 cc saline physiological saline will be applied to the subtenon space. 2nd group of patients (45 volunteers) will undergo a subtenon injection of Wharton gel-derived mesenchymal stem cell suspension. A suspension containing mesenchymal stem cell exosomes from Wharton jelly will be applied to the subtenon distance to the 3rd group of patients (45 volunteers). A single eye of each volunteer will be included. Informed consent will be obtained from the volunteers.

Allogeneic human Wharton gel tissue-derived mesenchymal stem cells and their exosomes will be obtained from healthy female volunteers, who is over 18 years old, under sterile conditions after HBV, HCV, HIV virus and "Treponema Pallidum" (VDRL) tests were performed. Cord tissue obtained from birth will be carried in a sterile transfer solution and will be processed to obtain stem cells in Erciyes University Genome and Stem Cell GMP (good manufacturing practices) certified laboratories. Exosomes will be obtained by the ultracentrifugation method in the same facility.

For injection into the subtenon distance, the conjunctiva and tenon will be opened with a small incision about 10 mm away from the lower temporal area, then 20 gauge curved subtenon cannula will be advanced parallel to the sclera and injected into the posterior subtenon area. All volunteers will be prescribed antibiotics and steroid drops after the surgical procedure.

Full ophthalmological examination and examinations at the beginning of the study will be performed and recorded again on the 1st day, 1st month, 2nd month, 3rd month and 6th months of the anterior segment and fundus examination, OCT (optical coherence tomography), VF (visual field) ), ERG (electroretinogram), mfERG (multifocal ERG), OCTA (optical coherence tomography) examinations will be performed.

In addition, a questionnaire evaluating the visual functions subjectively will be administered at the 1st, 3rd and 6th-month visits. (National Eye Institute Visual Functioning Questionnaire - 25 / National Eye Institute (USA) Visual Function Questionnaire ). Two masked investigators will perform analyses.

Post-procedure 1st Day, 1st Month, 2nd Month, 3rd Month and 6th Month data will be compared among study groups and within groups.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over,
* Diagnosis of retinitis pigmentosa: by clinical history, fundus examination, visual field (GA), electroretinogram (ERG), and genetic analysis
* Visual field loss
* The best corrected visual acuity of 0.05 on the Snellen chart
* The MD (mean deviation) value in the visual field is between 33.0 and -5.0 dB
* Intraocular pressure value below 22 mmHg

Exclusion Criteria:

* Presence of cataracts or other media opacities that may affect imaging and tests
* Diagnosis of glaucoma
* History of ocular surgery or injection in the last 6 months
* Visual level too low for examinations (0.05 and below)
* Diagnosis of any systemic disease (such as diabetes, uncontrolled hypertension, neurological disease)
* Smoking and substance abuse

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of best corrected visual acuity change | Upto 6 months
  Visual acuity change with LogMar Chart
Evaluation of visual field change | Upto 6 months
  Mean deviation values of automatic visual field testing

SECONDARY OUTCOMES:
Evaluation of multifocal ERG changes | Upto 6 months
  Amplitudes changes in multifocal ERG testing
Evaluation of ERG changes | Upto 6 months
  Amplitude changes in multifocal ERG testing
Evaluation of optical coherence tomography changes | Upto 6 months
  Retinal thickness changes in optical coherence tomography change
Evaluation of optical coherence tomography angiography changes | Upto 6 months
  Vascular density changes in optical coherence tomography angiography

CONTACTS AND LOCATIONS:
Overall Officials: Kuddusi ERKILIÇ, Professor, Principal Investigator — Erciyes University Medical Faculty
Locations (1):
- Erciyes University, Faculty of Medicine, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Limoli PG, Limoli CSS, Morales MU, Vingolo EM. Mesenchymal stem cell surgery, rescue and regeneration in retinitis pigmentosa: clinical and rehabilitative prognostic aspects. Restor Neurol Neurosci. 2020;38(3):223-237. doi: 10.3233/RNN-190970. PMID 32310198
- [Background] Bhattacharya S, Gangaraju R, Chaum E. Recent Advances in Retinal Stem Cell Therapy. Curr Mol Biol Rep. 2017 Sep;3(3):172-182. doi: 10.1007/s40610-017-0069-3. Epub 2017 Jul 10. PMID 29152454
- [Background] Limoli PG, Vingolo EM, Limoli C, Nebbioso M. Stem Cell Surgery and Growth Factors in Retinitis Pigmentosa Patients: Pilot Study after Literature Review. Biomedicines. 2019 Nov 30;7(4):94. doi: 10.3390/biomedicines7040094. PMID 31801246
- [Background] Borkowska-Kuczkowska A, Slugocka D, Swiatkowska-Flis B, Boruczkowski D. The use of mesenchymal stem cells for the treatment of progressive retinal diseases: a review. Regen Med. 2019 May;14(4):321-329. doi: 10.2217/rme-2019-0022. Epub 2019 Apr 12. PMID 30977436
- [Background] Jin ZB, Gao ML, Deng WL, Wu KC, Sugita S, Mandai M, Takahashi M. Stemming retinal regeneration with pluripotent stem cells. Prog Retin Eye Res. 2019 Mar;69:38-56. doi: 10.1016/j.preteyeres.2018.11.003. Epub 2018 Nov 9. PMID 30419340
- [Background] Ozmert E, Arslan U. Management of retinitis pigmentosa by Wharton's jelly derived mesenchymal stem cells: preliminary clinical results. Stem Cell Res Ther. 2020 Jan 13;11(1):25. doi: 10.1186/s13287-020-1549-6. PMID 31931872
- [Background] Oner A. Stem Cell Treatment in Retinal Diseases: Recent Developments. Turk J Ophthalmol. 2018 Feb;48(1):33-38. doi: 10.4274/tjo.89972. Epub 2018 Feb 23. PMID 29576896
- [Background] Cotrim CC, Jorge R, Oliveira MC, Pieroni F, Messias AMV, Siqueira RC. Clinical studies using stem cells for treatment of retinal diseases: state of the art. Arq Bras Oftalmol. 2020 Mar-Apr;83(2):160-167. doi: 10.5935/0004-2749.20200037. PMID 32159599
- [Background] Huo DM, Dong FT, Yu WH, Gao F. Differentiation of mesenchymal stem cell in the microenviroment of retinitis pigmentosa. Int J Ophthalmol. 2010;3(3):216-9. doi: 10.3980/j.issn.2222-3959.2010.03.08. Epub 2010 Sep 18. PMID 22553557
- [Background] Satarian L, Nourinia R, Safi S, Kanavi MR, Jarughi N, Daftarian N, Arab L, Aghdami N, Ahmadieh H, Baharvand H. Intravitreal Injection of Bone Marrow Mesenchymal Stem Cells in Patients with Advanced Retinitis Pigmentosa; a Safety Study. J Ophthalmic Vis Res. 2017 Jan-Mar;12(1):58-64. doi: 10.4103/2008-322X.200164. PMID 28299008
- [Background] Kuriyan AE, Albini TA, Townsend JH, Rodriguez M, Pandya HK, Leonard RE 2nd, Parrott MB, Rosenfeld PJ, Flynn HW Jr, Goldberg JL. Vision Loss after Intravitreal Injection of Autologous "Stem Cells" for AMD. N Engl J Med. 2017 Mar 16;376(11):1047-1053. doi: 10.1056/NEJMoa1609583. PMID 28296617
- [Background] Harrell CR, Fellabaum C, Jovicic N, Djonov V, Arsenijevic N, Volarevic V. Molecular Mechanisms Responsible for Therapeutic Potential of Mesenchymal Stem Cell-Derived Secretome. Cells. 2019 May 16;8(5):467. doi: 10.3390/cells8050467. PMID 31100966
- [Background] Klingeborn M, Dismuke WM, Bowes Rickman C, Stamer WD. Roles of exosomes in the normal and diseased eye. Prog Retin Eye Res. 2017 Jul;59:158-177. doi: 10.1016/j.preteyeres.2017.04.004. Epub 2017 Apr 29. PMID 28465248
- [Background] Harrell CR, Simovic Markovic B, Fellabaum C, Arsenijevic A, Djonov V, Arsenijevic N, Volarevic V. Therapeutic Potential of Mesenchymal Stem Cell-Derived Exosomes in the Treatment of Eye Diseases. Adv Exp Med Biol. 2018;1089:47-57. doi: 10.1007/5584_2018_219. PMID 29774506
- [Background] Mead B, Tomarev S. Extracellular vesicle therapy for retinal diseases. Prog Retin Eye Res. 2020 Nov;79:100849. doi: 10.1016/j.preteyeres.2020.100849. Epub 2020 Mar 10. PMID 32169632
- [Background] Yaghoubi Y, Movassaghpour A, Zamani M, Talebi M, Mehdizadeh A, Yousefi M. Human umbilical cord mesenchymal stem cells derived-exosomes in diseases treatment. Life Sci. 2019 Sep 15;233:116733. doi: 10.1016/j.lfs.2019.116733. Epub 2019 Aug 5. PMID 31394127
- [Background] Zhang X, Liu J, Yu B, Ma F, Ren X, Li X. Effects of mesenchymal stem cells and their exosomes on the healing of large and refractory macular holes. Graefes Arch Clin Exp Ophthalmol. 2018 Nov;256(11):2041-2052. doi: 10.1007/s00417-018-4097-3. Epub 2018 Aug 30. PMID 30167916
- [Background] Ma M, Li B, Zhang M, Zhou L, Yang F, Ma F, Shao H, Li Q, Li X, Zhang X. Therapeutic effects of mesenchymal stem cell-derived exosomes on retinal detachment. Exp Eye Res. 2020 Feb;191:107899. doi: 10.1016/j.exer.2019.107899. Epub 2019 Dec 19. PMID 31866431
- [Background] Yu B, Shao H, Su C, Jiang Y, Chen X, Bai L, Zhang Y, Li Q, Zhang X, Li X. Exosomes derived from MSCs ameliorate retinal laser injury partially by inhibition of MCP-1. Sci Rep. 2016 Sep 30;6:34562. doi: 10.1038/srep34562. PMID 27686625
- [Background] Zhang W, Wang Y, Kong Y. Exosomes Derived From Mesenchymal Stem Cells Modulate miR-126 to Ameliorate Hyperglycemia-Induced Retinal Inflammation Via Targeting HMGB1. Invest Ophthalmol Vis Sci. 2019 Jan 2;60(1):294-303. doi: 10.1167/iovs.18-25617. PMID 30657854
- [Background] Hajrasouliha AR, Jiang G, Lu Q, Lu H, Kaplan HJ, Zhang HG, Shao H. Exosomes from retinal astrocytes contain antiangiogenic components that inhibit laser-induced choroidal neovascularization. J Biol Chem. 2013 Sep 27;288(39):28058-67. doi: 10.1074/jbc.M113.470765. Epub 2013 Aug 7. PMID 23926109
- [Background] Ha DH, Kim SD, Lee J, Kwon HH, Park GH, Yang SH, Jung JY, Lee JH, Park SR, Youn J, Lee SH, Kim JE, Lim J, Lee HK, Cho BS, Yi YW. Toxicological evaluation of exosomes derived from human adipose tissue-derived mesenchymal stem/stromal cells. Regul Toxicol Pharmacol. 2020 Aug;115:104686. doi: 10.1016/j.yrtph.2020.104686. Epub 2020 May 22. PMID 32450131
- [Background] Pan D, Chang X, Xu M, Zhang M, Zhang S, Wang Y, Luo X, Xu J, Yang X, Sun X. UMSC-derived exosomes promote retinal ganglion cells survival in a rat model of optic nerve crush. J Chem Neuroanat. 2019 Mar;96:134-139. doi: 10.1016/j.jchemneu.2019.01.006. Epub 2019 Jan 10. PMID 30639447
- [Background] Zhao T, Liang Q, Meng X, Duan P, Wang F, Li S, Liu Y, Yin ZQ. Intravenous Infusion of Umbilical Cord Mesenchymal Stem Cells Maintains and Partially Improves Visual Function in Patients with Advanced Retinitis Pigmentosa. Stem Cells Dev. 2020 Aug;29(16):1029-1037. doi: 10.1089/scd.2020.0037. Epub 2020 Jul 15. PMID 32679004